CLINICAL TRIAL: NCT00230360
Title: Diagnosis of Functional Defecation Disorders in Childhood
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Other Study IDs: AU-20050020
Record Dates: First submitted 2005-09-29; First posted 2005-09-30 (Estimated); Last update posted 2007-02-02 (Estimated); Status verified 2007-02

CONDITIONS: Constipation; Fecal Incontinence
Keywords: constipation; fecal incontinence; diagnosis; children
MeSH Terms: conditions — Constipation; Fecal Incontinence; Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Purpose To compare different kinds of diagnostic investigations in order to identify the most sensitive and least invasive when diagnosing constipation.

DETAILED DESCRIPTION:
Defecation disorders in children are extremely common especially constipation and fecal incontinence. International studies show that constipation make up approximately 3% of Pediatric Outpatient Clinic11 (192) and 25% of Pediatric gastroenterology consultations. Between 1,5-3% of all 4-12 year olds experience fecal incontinence.

Constipation and fecal incontinence can be extremely physical unpleasant and can have significant ramifications for a child's emotional and social functioning eg. low self esteem.

Though most agree that constipation and faecal incontinence are a considerable problem worldwide there is disagreement when it comes to a definition and diagnostic tools. Several definitions have been used. This has led to great difficulties when trying to estimate prevalence, understand and compare in order to improve different treatments.

Hypothesis:

* It is possible to diagnose constipation accurately by using a combination of anamnesis, stool diary, physical examination and transabdominal ultrasonography
* Transabdominal ultrasonography is a safe and sensitive diagnostic tool and can be used as an alternative or substitute to rectal examination.

Purpose To compare different kinds of diagnostic (tools) investigations in order to identify the most sensitive and least invasive when diagnosing constipation.

Material and methods 60 children referred to the paediatric outpatient clinic with fecal incontinence or suspicion of constipation. The investigations include anamnesis and physical examination with rectal examination and transabdominal ultrasonography. Home registration of a stool diary based on the Bristol Scale for 3 weeks thereafter a Colonic transit time is performed.

Data is compared to data from 30 healthy children that have gone through the same investigations except the CTT that is based on x-rays.

ELIGIBILITY:
Inclusion Criteria:

Referred children

* functional constipation and/or fecal incontinence

Healthy children

* No sign of functional constipation and/or fecal incontinence

Exclusion Criteria:

Referred children

* organic constipation/ fecal incontinence

Healthy children

* constipation/ fecal incontinence

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90
Dates: Start 2005-06; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Overall Officials: Iben M Jonsson, Med Student, Principal Investigator — University of Aarhus; Soren Rittig, MD, Study Director — University of Aarhus
Locations (1):
- Department of Pediatrics, Aarhus University Hospital, Skejby Sygehus, Aarhus, Denmark